CLINICAL TRIAL: NCT05613660
Title: A Proof of Science Clinical Study With Randomized, Four Arm, Comparative, Single-Blind, Within the Arm - Dose-Response Study to Evaluate the Safety, Efficacy of Different Collagen Peptide Containing Test Treatments in Adult Human Subjects
Brief Title: A Proof of Science, Dose-Response Study to Evaluate the Safety, Efficacy of Different Dosages of Test Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Collagen Lifesciences Private Limited (Unknown)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator - Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NB220031-COL
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Mild to Moderate Acne; Stiffness of Joint, Nec, Involving Ankle and Foot in MDR24_1; Other Specified Diseases of Hair and Hair Follicles; Brittle Nails; Osteoarthritis, Knee; Healthy
Keywords: Acne, Wrinkles, Joints pain, brittle nails, hair fall
MeSH Terms: conditions — Enterocolitis, Necrotizing; Twenty-Nail Dystrophy; Osteoarthritis, Knee; Acne Vulgaris; Arthralgia

STUDY DESIGN:
Intervention Model Description: Proof of Science, Randomized, Four-arm, Comparative, Single-Blind, Evaluator-Blinded, Dose Response, Safety and Efficacy Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned in as 1:1:1:1 ratio to receive either treatment A or B or C or D and three different dosages i.e. 2.5g, 5g, and 10g. The randomization code will be generated by NovoBliss Research. Single-blind will be followed for the evaluators.
  Subjects will be randomly allocated to one of the treatment groups and one of treatment dose, as per the randomization code. This is single-blind study and blinding will be kept wherein neither the evaluator staff nor the Investigator shall be aware of the test treatment or test treatment dose allocation (except for osteoarthritis patients for Bovine Test Treatment). To maintain blinding, the study staff who involves in treatment dispensing and distribution will not be involved in any other study-related activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VEGCOL™️ (Veg Collagen Peptide) (Experimental): Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water
  VEGCOL helps in providing the necessary nutrition needed for the body to produce collagen. Vegan collagen gives a lighter feel on consumption compared to any other collagen and increases the elasticity of the skin and makes skin supple. VEGCOL has more amino acids than animal derived Collagen which makes it very ideal to consume not only in Vegetarian populated countries like in India but around the world. Pepsin, a digestive enzyme, is added to help structure the building blocks into collagen molecules with the exact structure of human collagen.
  Interventions: Dietary Supplement: Veg Collagen Peptide
- PROCOL (Bovine Collagen Peptide) (Experimental): Bovine collagen is a naturally occurring protein present in the connective tissue, bones, cartilage, and hides of cows.
  Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water.
  Interventions: Dietary Supplement: Bovine Collagen Peptide
- AQUACOL (Fish | Marine Collagen Peptide) (Experimental): Marine Collagen is made from Fish Skin which delays the signs of aging such as wrinkles, Joint issues and weakness.
  Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water.
  Interventions: Dietary Supplement: Fish | Marine Collagen Peptide
- CALCOL (Chicken Collagen Peptide) (Experimental): Chicken collagen is used to treat joint pain associated with many types of arthritis and surgery, as well as back pain, neck pain, and pain following injury. Chicken collagen works by causing participants' body to produce substances that fight inflammation and pain. It also contains chondroitin and glucosamine, two compounds that help rebuild cartilage. That's why chicken collagen can provide some amazing benefits for participants' gut, immune system, skin, and more.
  Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water.
  Interventions: Dietary Supplement: Chicken Collagen Peptide

INTERVENTIONS:
Dietary Supplement: Veg Collagen Peptide — Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water
  Other Names: VEGCOL™️
  Arms: VEGCOL™️ (Veg Collagen Peptide)
Dietary Supplement: Bovine Collagen Peptide — Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water
  Other Names: PROCOL
  Arms: PROCOL (Bovine Collagen Peptide)
Dietary Supplement: Fish | Marine Collagen Peptide — Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water
  Other Names: AQUACOL
  Arms: AQUACOL (Fish | Marine Collagen Peptide)
Dietary Supplement: Chicken Collagen Peptide — Mode of Usage: 1 scoop/sachet daily Route of Administration: Oral administration with a glassful (approx. 250 mL) of water
  Other Names: CALCOL
  Arms: CALCOL (Chicken Collagen Peptide)

SUMMARY:
A proof of science clinical study with randomized, four-arm, comparative, single-blind, within the arm - Dose-Response Study to evaluate the safety and efficacy of different collagen peptide-containing test treatments in adult human subjects.

The dose-response will be evaluated for the effectiveness of each test treatment in three different dosages that is 2.5 g Versus 5 g Versus 10 g.

22 subjects will be enrolled per dose per test treatment to complete 20 subjects per dose per test treatment.

DETAILED DESCRIPTION:
A proof of science clinical study with randomized, four-arm, comparative, single-blind, within the arm - Dose-Response Study to evaluate the safety and efficacy of different collagen peptide-containing test treatments in adult human subjects.

The dose response will be evaluated for the effectiveness of each test treatment in three different dosages that is 2.5 g Versus 5 g Versus 10 g.

22 subjects will be enrolled per dose per test treatment to complete 20 subjects per dose per test treatment.

There are four different test treatments as mentioned below will be tested during study.

* Test Treatment A: VEGCOL™️ (Veg Collagen Peptide)
* Test Treatment B: PROCOL (Bovine Collagen Peptide)
* Test Treatment C: AQUACOL (Fish/Marine Collagen Peptide)
* Test Treatment D: CALCOL (Chicken Collagen Peptide) Mode of Usage: 1 scoop/sachet of daily Route of Administration: Oral Administration with a glassful (approx. 250 mL) of water.

Considering proof of science study, a sufficient number of adult subjects with an age group of 30 - 50 years old (i) having mild to moderate crows' feet wrinkles near to eye area and (ii) mild to moderate joints pain, swelling, stiffness and decreased range of motion (iii) having complaints of hair fall, decreased hair growth, brittle nails will be recruited/enrolled.

In Bovine Arm, out of 66 subjects, a few subjects with osteoarthritis patients having present complaints of pain and stiffness in joints will be enrolled.

The collagen peptides effects of all 4 variants will be evaluated in enrolled subjects with mild to moderate acne.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day -04): Screening, Baseline evaluations
* Visit 02 (Day 01): Enrolment, Hair Growth Rate measurement, Evaluations
* Visit 03 (Day 10): Treatment Period, Evaluations
* Visit 04 (Day 30): Treatment Period, Evaluations
* Visit 05 (Day 57): Treatment Period, Evaluations, Tattoo, Hair growth measurement
* Visit 06 (Day 60): Evaluations, End of Study Visit

Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be telephonically contacted by recruiting department prior to the enrolment visit. Subjects will be instructed during screening (prior to enrolment) not to wear any facial makeup during study visits to the facility. The study will be conducted in four different groups considering four different arms of test treatments.

Assessment of safety and efficacy parameters will be done before test treatment usage on Day 1, and will be compared with after test treatments usage on Day 10 (+2 Days), Day 30 (+2 Days), and Day 60 (+2 Days) within treatments and between treatments, between three dosages as listed-below.

* Skin Elasticity: DermaLab®Combo (Right cheek)
* Deep Skin Hydration: MoitureMeterEPiD (Right cheek)
* Skin Moisture for Skin Barrier Function: Vapometer (Right Cheek)
* Crow's feet area wrinkles, fine lines, skin texture - roughness, dryness, wrinkles, smoothness: Visioscan (C+K Instrument)
* Improvement in Glogau Skin Age : Dermatological evaluation
* Improvement in PGA Dermatologist Scoring using Griffiths Scale - Skin dryness, redness, fine wrinkles/lines, coarse wrinkling/lines, laxity, roughness, and sallowness : Dermatological evaluation
* Change of the PGA score for assessment of the signs of brittle nails
* Change of the PGA score for assessment of Acne
* Hair Strength: Hair Pull test
* Hair Fall Reduction: 60-second hair count (Hair Combing Method)
* Hair Growth, Thickness, Density: CASLite Nova (Phototrichogram)
* A:T Ratio (Hair Growth Cycle): Pluck Test - Trichogram (Microscopic Evaluation)
* Hight, Weight, BMI - Anthropometry
* Leeds Sleep Evaluation Questionnaire (LSEQ) - Deep and Sound Sleep
* Hedonic Questionnaires - about product perception and consumer feedback. - Skin elasticity, suppleness, deep and sound sleep, digestion and gut health, joint health, nail, and hair health
* Change in Pain According to VAS (0-10 cm) for arthritis complaints
* Consumption of Rescue Medication for osteoarthritis patients/subjects
* Change in muscles strength - as assessed by the sum of the handgrip, elbow flexion and extension, and knee flexion and extension strength by the dynamometer
* Digital Photographs: Facial photographs [Left, Center, Right] and Nails photographs before test treatment usage and after test treatment usage.

ELIGIBILITY:
Inclusion Criteria:

The subject must fulfil all of the following inclusion criteria to be eligible for participation in the study unless otherwise specified.

1. Age: 30 to 50 years (both inclusive) at the time of consent.
2. Sex: Healthy non-pregnant/non-lactating females and Males.
3. Female of childbearing potential must have a reported negative pregnancy during screening and end of the study.
4. Subject is generally in good health.
5. Subject has mild to moderate crows' feet wrinkles.
6. Subject has mild to moderate joints pain, swelling, stiffness and decreased range of motion.
7. Subject has a score of at least "mild skin aging" based on PGA at screening visit.
8. Subject has Glogau Skin Age II or III as assessed by the Dermatologist/ Dermatologist Trained Evaluator.
9. Subject having complaints of hair fall and decreased hair growth.
10. The subject self-declare nonpathological thin, dry, and brittle hair and nails.
11. Subject is willing to forgo cosmetic procedures 3 months prior to and for the duration of the study.
12. Subject is able to follow their normal skin care routines and to refrain from introducing any new skin care products during the study.
13. Subject is able to forgo changes in baseline medications and nutritional supplements, any other collagen peptide powder during the study period.
14. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
15. If the female subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
16. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
17. Subject is willing not to introduce any new soaps, cleansers, lotions, creams, or any other face product etc. for the duration of the study.
18. Subject is willing to give written informed consent and are willing to follow the study procedure.
19. Subject is committed not to not to use medicated/ prescription shampoos/hair care products (containing Minoxidil / Anti-thinning agents) or any other hair growth, treatment for thin hair, or hair products other than the test product for the entire duration of the study.
20. The subject is willing to use test treatment throughout the study period.
21. Only For Bovine Arm: Subjects with osteoarthritis patients having present complaints of pain and stiffness in joints (based on their current prescription and medical history).

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any one of the following criteria:

1. Subject has a history of allergy or sensitivity to the test treatments ingredients.
2. Subject who has a history of allergy with products containing Fish, Bovine, Chicken, broccoli and carrots.
3. Subject who has pre-existing or dormant dermatologic conditions (e.g., psoriasis rashes, eczema, seborrheic dermatitis, acne or any other) that could interfere with the outcome of the study as determined by the Investigator.
4. Subject has used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
5. Subject has applied any topical retinoids within 2 weeks of the screening visit or anticipates having to use at any point during the study.
6. Subject is not willing to avoid unprotected sun or other UV radiation exposure during the study period.
7. Subject has a history of prior use of hair growth treatment within 3 months.
8. Subject has a history of any prior hair growth procedures (e.g., hair transplant or laser).
9. Subject has a history of alcohol or drug addiction.
10. Subject has plans of shaving scalp hair during the study.
11. Subject is currently participating in or planning on starting a weight loss program that may result in a significant change in overall body weight.
12. Subject has a history of prior use of skin radiance or wrinkle laser treatment within 3 months.
13. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
14. Pregnant or breastfeeding or planning to become pregnant during the study period.
15. Subject has a history of chronic illness which may influence the cutaneous state.
16. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials or skin care products within the last four weeks

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the facial wrinkles and fine lines of Crow's feet area, skin texture - roughness, dryness, wrinkles, smoothness | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in the facial wrinkles and fine lines of Crow's feet area, skin texture - roughness, dryness, wrinkles, smoothness using Visioscan® VC 20 Plus after 8 weeks of treatment, between treatments, between three different dosages and within a treatment
Change in Skin Elasticity | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments in skin elasticity using DermaLab®Combo or equivalent (Right cheek) after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in Skin Hydration | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments in skin hydration using MoitureMeterEPiD (Right cheek) after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in Hair Thickness and Density | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Hair Thickness and Density in using CASLiteNova through Phototrichogram after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in Hair Fall | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in hair fall using a 60-second hair count (Hair Combing Method) after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in Body Weight and BMI | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in body weight in Kg and Body Mass Index (BMI) Kg/m2 after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in Joints Pain using VAS (0-10 cm) scoring evaluated by trained study staff | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Joints Pain using VAS (0-10 cm) scoring evaluated by trained study staff after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
Change in muscles strength | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in muscle strength as assessed by the sum of the handgrip, elbow flexion, and extension, and knee flexion and extension strength evaluated by trained study staff after 8 weeks of treatment, between treatments, between three different dosages, and within a treatment
To assess the effect of test treatment in terms of change in hair growth on the scalp | Baseline visit i.e. during Visit 01 (04 days before Day 01) and Visit 02 (Day01) before application to Visit 05 (Day 57) and Visit 06 (Day 60)
  Hair growth rate (µm/day) will be measured by using data of hair growth from Visit 01 and Visit 02 for baseline reading and from Visit 05 and Visit 06 for post-treatment reading.
  Note: Hair growth rate (μm/day) will be measured by using data of hair growth from Visit 01 and Visit 02 for baseline reading and from Visit 05 and Visit 06 for post-treatment reading

SECONDARY OUTCOMES:
Change in Physician Global Assessment (PGA) scoring - Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Physician Global Assessment (PGA) scoring using the Griffiths scale - Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness after 8 weeks of treatment, between treatments, between three different dosages and within the treatment evaluated by dermatologist trained scorer
Change in Glogau Skin Age | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Glogau Skin Age after 8 weeks of treatment, between treatments, between three different dosages and within the treatment evaluated by a dermatologist trained scorer
Change on hair strength by Pull test | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in scalp hair strength using the pull test method evaluated by dermatologist-trained scorer after 8 weeks of treatment, between treatments, between three different dosages, and within the treatment
Change in Physician Global Assessment (PGA) score for assessment of the signs of brittle nails, surface roughness, raggedness, and peeling | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Physician Global Assessment (PGA) score for assessment of the signs of brittle nails, surface roughness, raggedness, and peeling evaluated by dermatologist-trained scorer after 8 weeks of treatment, between treatments, between three different dosages, and within the treatment
Change in Sleep Quality using Leeds Sleep Evaluation Questionnaires (LSEQ) | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in Sleep Quality using Leeds Sleep Evaluation Questionnaires (LSEQ) evaluated by trained staff after 8 weeks of treatment, between treatments, between three different dosages, and within the treatment
Consumption of Rescue Medications for Joints pain | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for the requirement of consumption of rescue medications for Joints pain during and after 8 weeks of treatment, between treatments, between three different dosages, and within the treatment
Test treatment perception and consumer feedback on Skin elasticity, suppleness, deep and sound sleep, digestion and gut health, joint health, and nail and hair health | Baseline (Day01) to Day 10 (+2Days), Day 30 (+2Days) and Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments perception and consumer feedback on skin elasticity, suppleness, deep and sound sleep, digestion and gut health, joint health, and nail and hair health using hedonic questionnaires evaluated by trained study staff after 8 weeks of treatment, between treatments, between three different dosages, and within the treatment
Change in Physician Global Assessment (PGA) score for assessment of Acne Severity | Baseline (Day01) to Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments for change in PGA score of acne severity evaluated by dermatologist trained scorer in enrolled subjects with mild to moderate acne - between treatments, between three different dosages, and within the treatment
Change in Anagen Telogen (A:T) ratio | Baseline (Day01) to Day 60 (+2Days)
  To evaluate the effectiveness of the test treatments after 8 weeks of treatment in Anagen Telogen (A:T) ratio using pluck test - between treatments, between three different dosages and within treatment evaluated by dermatologist trained scorer to assess Hair growth cycle (Trichogram)
Change in facial photographs (left/center/right) and nails photographs of the subjects | Baseline (Day01) to Day 60 (+2Days)
  Change in facial photographs (left/center/right) and nails photographs of the subjects in three different dosages and between treatments will be presented at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No